CLINICAL TRIAL: NCT01016743
Title: The Influence of Low Frequency Repetitive Transcranial Stimulation (r-TMS) on Motor and Cognitive Measurements in Patients With Asymmetric Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sheba Medical Center: Dr. Oren Cohen PI, Sheba Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-09-7279-OC-CTIL
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: UPDRS
Keywords: parkinson; rTMS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active repetitive transcranial Stimulation (Active Comparator): Patients will be randomized into two groups: The first group of patients will receive an active unilateral stimulation over the motor cortex contralateral to the more affected body side (1Hz stimulation 110% of the MT for 15 minutes). Patients in the second group will receive a similar rTMS stimulation pattern over the motor cortex and over the prefrontal cortex (10Hz stimulation 100% of the MT, 2 seconds each train, 20 seconds between trains, for 15 minutes).
  Interventions: Device: repetitive transcranial stimulation (r-TMS)

INTERVENTIONS:
Device: repetitive transcranial stimulation (r-TMS) — Patients will be randomized into two groups: The first group of patients will receive an active unilateral stimulation over the motor cortex contralateral to the more affected body side (1Hz stimulation 110% of the MT for 15 minutes). Patients in the second group will receive a similar rTMS stimulation pattern over the motor cortex and over the prefrontal cortex (10Hz stimulation 100% of the MT, 2 seconds each train, 20 seconds between trains, for 15 minutes).

SUMMARY:
To test the effects of low frequency deep rTMS using the novel H-coil on the motor, affective and cognitive deficits in patients with asymmetric Parkinson's disease (PD) and to establish its safety in this population. The investigators anticipate that reaching deeper brain layers and larger volume of activation with the novel H-coil may induce significantly better therapeutic effects in patients with PD and will pave the way for establishing a novel and effective treatment for this disorder.

DETAILED DESCRIPTION:
PD patients with asymmetric disease aged 40 years or older, diagnosed as idiopathic PD according to the UK Brain Bank criteria, with Hoehn & Yahr stages II - IV while "off" will be recruited. Participants on antidepressants should be at least 2 months on stable therapy.

Patient will be excluded if:

1. They have concomitant epilepsy, a history of seizure or heat convulsion or history of epilepsy in first degree relative.
2. Are on neuroleptics.
3. Have dementia or any unstable medical disorder.
4. Have a history or current unstable hypertension.
5. Have a history of head injury or neurosurgical interventions.
6. Have a history of any metal in the head (outside the mouth).
7. Have a known history of any metallic particles in the eye, implanted cardiac pacemaker, implanted neurostimulators, surgical clips (above the shoulder line) or any medical pumps.

Patients will be randomized into two groups: The first group of patients will receive an active unilateral stimulation over the motor cortex contralateral to the more affected body side (1Hz stimulation 110% of the MT for 15 minutes). Patients in the second group will receive a similar rTMS stimulation pattern over the motor cortex and over the prefrontal cortex (10Hz stimulation 100% of the MT, 2 seconds each train, 20 seconds between trains, for 15 minutes).

The following outcome measures will be taken prior to the treatment (screening visit), and at day 1, 10, 30 and 60 Evaluation will be while subjects both at "on" and "off".

Motor:

1. Unified Parkinson's Disease Rating Scale (UPDRS )
2. Clinical Global Impression of Severity (CGIS)
3. Pegboard test.
4. Tapping test
5. Up & Go test
6. Abnormal Involuntary Movement Scale (AIMS) Mood and affect

1. Beck Depression Inventory (BDI) Cognition

1. Mini mental State examination (MMSE)
2. Digit forward and backward tests.
3. Word fluency.
4. Frontal Assessment Battery (FAB) Side effects will be closely monitored by the researchers and will be promptly reported to the IRB.

8.Have a history of migraine or frequent or severe headaches. 9.Have a history of hearing loss. 10.Has a of cochlear implants 11.Have a history of drug abuse or alcoholism. 12.Is pregnant or not using a reliable method of birth control. 13.Is participating in current clinical study or clinical study within 30 days prior to this study.

ELIGIBILITY:
Inclusion Criteria:

* PD patients with asymmetric disease aged 40 years or older, diagnosed as idiopathic PD according to the UK Brain Bank criteria, with Hoehn & Yahr stages II - IV while "off".
* Participants on antidepressants should be at least 2 months on stable therapy.

Exclusion Criteria:

* Patients who have concomitant epilepsy, a history of seizure or heat convulsion or history of epilepsy in first degree relative.
* Patients on neuroleptics.
* Patients with dementia or any unstable medical disorder.
* History or current unstable hypertension.
* History of head injury or neurosurgical interventions.
* History of any metal in the head (outside the mouth).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS ) | 1 year

SECONDARY OUTCOMES:
CGIS,Pegboard test.Tapping test,Up&Go test,AIMS,BDI,MMSE,Word fluencyFAB | 1 year
UPDRS | 3 months